CLINICAL TRIAL: NCT06766890
Title: Evaluation of Innovative School-based Interventions on Health Outcomes Among Primary School Students During Post COVID-19 Pandemic
Acronym: WeJoy+WeHop
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lau Ying, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CV-2024-YL
Record Dates: First submitted 2024-12-31; First posted 2025-01-09 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Childhood Obesity; Sleep Problems; Physical Activity
Keywords: Innovative school-based intervention; School children; Cognitive behavioral therapy; Exergaming
MeSH Terms: conditions — Pediatric Obesity; Parasomnias; Motor Activity

STUDY DESIGN:
Intervention Model Description: 1:1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- School-based Cognitive Behavior Therapy (WeJoy and exergaming on the interactive floor (WeHop) (Experimental): School-based CBT (WeJoy) allows children to recognize, change, and partake in pleasant activities based on the CBT model. The WeJoy comprises six weekly sessions on psychoeducation, cognitive restructuring, behavioural activation, emotional regulation, and self-monitoring. Exergaming on the interactive floor (WeHop) using a portable interactive projector games system. Each session provides 2 to 3 games per week for six weeks.
  Interventions: Behavioral: WeJoy+WeHop
- Usual class (No Intervention): Usual extra curriculum activities that are arranged by corresponding primary schools

INTERVENTIONS:
Behavioral: WeJoy+WeHop — School-based CBT (WeJoy) comprises six weekly sessions on psychoeducation, cognitive restructuring, behavioural activation, emotional regulation, and self-monitoring. Exergaming on the interactive floor (WeHop) can gain a sense of autonomy, competence, and relatedness to help them regulate their emotions and maintain positive behaviours according to the Self-Determination Theory. Children participate in the interactive floor games by stepping on various targets and moving in response to the game's rules. Combining task division, cooperation, and taking turns constitutes the collaboration mechanism.
  Arms: School-based Cognitive Behavior Therapy (WeJoy and exergaming on the interactive floor (WeHop)

SUMMARY:
Objectives: (1) to evaluate the feasibility of innovative school-based interventions on health outcomes (psychological well-being, depressive symptoms, anxiety symptoms, physical activity, sleep duration, and sleep quality) among primary students in the post-COVID-19 pandemic period; (2) to explore children's experience of intervention; (3) to evaluate the effects of innovative school-based (WeJoy + WeHop) on depressive symptoms, physical activities, and sleep quality among primary 3 to 5 school children.

Method: Two phases of the study will be conducted, including feasibility pilot study and main study. In phase 1, a sample of 40 school children will be recruited from two community centers for feasibility test and semi-structured individual face-to-face interview. In phase 2, a total of 408 school children will be recruited from primary schools in Hong Kong. This study will adopt a 2 two-group pre and post-design. Participants are randomly assigned equally into 1 intervention group (WeJoy+WeHop) and 1 control group (Routine Extra curriculum Activity). Participants will be assessed at baseline and post-intervention. The outcomes are depressive symptoms, physical activities, and sleep quality, using the Chinese version of the Center for Epidemiologic Studies Depression Scale for Children (CES-DC), the Chinese Version of the International Physical Activity Questionnaire (IPAQ-C), and the Chinese version of the Pittsburgh Sleep Quality Index (PSQI-C).

Data analysis: Descriptive and inferential statistics will be performed to examine the research objectives.

DETAILED DESCRIPTION:
The COVID-19 pandemic has altered children's lifestyles, calling for particular attention. Psychological problems, obesity, and sleep disturbance in children have become more prevalent throughout the COVID-19 outbreak. It is vital to develop preventative interventions to enhance psychological well-being, prevent obesity, and improve sleep health. Cognitive behavioural therapy (CBT) is effective in preventing psychological problems, obesity, and sleep problems in children. The provision of CBT faces obstacles such as a shortage of therapists, stigma, protracted wait times, and high costs. Evidence revealed that children prefer interventions with interactive, relatable, and game-like content to improve their engagement.

School-based CBT (WeJoy) allows children to recognize, change, and partake in pleasant activities based on the CBT model. The WeJoy comprises six weekly sessions on psychoeducation, cognitive restructuring, behavioural activation, emotional regulation, and self-monitoring. Exergaming on the interactive floor (WeHop) using a portable interactive projector games system. The WeHop can gain a sense of autonomy, competence, and relatedness to help them regulate their emotions and maintain positive behaviours according to the Self-Determination Theory. Children participate in the interactive floor games by stepping on various targets and moving in response to the game's rules. Combining task division, cooperation, and taking turns constitutes the collaboration mechanism.

ELIGIBILITY:
Inclusion Criteria:

* Primary students ranged from primary 3 to 5 school children.
* Obtained consent forms from their legal guardians.

Exclusion Criteria:

* Primary students in primary 1 due to the adaptation of the new environment.
* Primary 6 due to the preparation of the examinations for secondary schools.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-02-23 (Actual); Primary Completion 2025-06-19 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Psychological outcome: Depressive symptoms | baseline, pre-intervention and immediately after the intervention
  Depressive symptoms will be assessed by the Chinese version of 20-item Center for Epidemiologic Studies Depression Scale for Children, CES-DC

SECONDARY OUTCOMES:
Physical activity | baseline, pre-intervention and immediately after the intervention
  Level of physical activities will be measured by the Chinese Version of 7-item International Physical Activity Questionnaire, IPAQ-C
Sleep outcomes include subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, sleep medication, and daytime dysfunction | baseline, pre-intervention and immediately after the intervention
  Subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, sleep medication, and daytime dysfunction will be assessed by the Chinese version of 19-item Pittsburgh Sleep Quality Index, Chinese PSQI

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
The data does not collect yet and the research team does not decide the plan to share IPD.